CLINICAL TRIAL: NCT03121482
Title: High-flow Nasal Cannula Oxygen Therapy With or Without Non-invasive Ventilation (NIV) During the Weaning Period: a Multicenter Randomized Controlled Trial
Brief Title: High-flow Nasal Cannula Oxygen Therapy With or Without NIV During the Weaning Period
Acronym: HIGH-WEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIGH-WEAN Study; 2016-A01078-43 (Other: CPP)
Record Dates: First submitted 2017-03-23; First posted 2017-04-20 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Acute Respiratory Failure Requiring Reintubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC alone (Active Comparator): Control group
  Interventions: Device: HFNC
- HFNC and NIV (Experimental)
  Interventions: Device: HFNC; Device: NIV

INTERVENTIONS:
Device: HFNC — Gas flow of 50 l/min and FiO2 adjusted to obtain SpO2 ≥ 92%
Device: NIV — Pressure-support level to achieve an expired tidal volume between 6 and 8 ml/kg and PEEP level of 5 cm H2O with FiO2 adjusted to obtain SpO2 ≥ 92%
  Arms: HFNC and NIV

SUMMARY:
Prospective multicenter randomized controlled open-label trial comparing 2 strategies of oxygenation during the post-extubation period in ICU patients at high risk of extubation failure. Patients will be randomized and assigned to one of the two groups, with a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Duration of mechanical ventilation prior to extubation at least 24h
* Planned extubation decided by the physician in charge of the patient after success of a weaning trial
* Patients at high risk of reintubation according to the following criteria: patients older than 65 years, or those having any underlying chronic cardiac or lung disease.

Exclusion Criteria:

* Patient admitted for traumatic brain injury
* Periphal neuromuscular disease as reason for intubation
* Usual lon-term treatment with NIV for chronic desease
* Usual lon-term treatment with CPAP for obstructive apneas syndrome
* Contraindication to NIV
* Unplanned extubation
* Do-not-reintubated order at time of extubation
* Terminal extubation for end of life
* People under legal protection
* Opposition to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Reintubation at Day 7 | up to 7 days
  The rate of reintubation will be assessed within the 7 days following planned extubation

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud W THILLE, Principal Investigator — CHU Poitiers
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thille AW, Coudroy R, Nay MA, Gacouin A, Decavele M, Sonneville R, Beloncle F, Girault C, Dangers L, Lautrette A, Levrat Q, Rouze A, Vivier E, Lascarrou JB, Ricard JD, Mekontso-Dessap A, Barberet G, Lebert C, Ehrmann S, Massri A, Bourenne J, Pradel G, Bailly P, Terzi N, Dellamonica J, Lacave G, Robert R, Frat JP, Ragot S; HIGH-WEAN Study Group and the REVA Research Network. Beneficial Effects of Noninvasive Ventilation after Extubation in Obese or Overweight Patients: A Post Hoc Analysis of a Randomized Clinical Trial. Am J Respir Crit Care Med. 2022 Feb 15;205(4):440-449. doi: 10.1164/rccm.202106-1452OC. PMID 34813391
- [Derived] Thille AW, Monseau G, Coudroy R, Nay MA, Gacouin A, Decavele M, Sonneville R, Beloncle F, Girault C, Dangers L, Lautrette A, Levrat Q, Rouze A, Vivier E, Lascarrou JB, Ricard JD, Razazi K, Barberet G, Lebert C, Ehrmann S, Massri A, Bourenne J, Pradel G, Bailly P, Terzi N, Dellamonica J, Lacave G, Robert R, Ragot S, Frat JP; HIGH-WEAN Study Group and the REVA research network. Non-invasive ventilation versus high-flow nasal oxygen for postextubation respiratory failure in ICU: a post-hoc analysis of a randomized clinical trial. Crit Care. 2021 Jun 28;25(1):221. doi: 10.1186/s13054-021-03621-6. PMID 34183053
- [Derived] Thille AW, Coudroy R, Nay MA, Gacouin A, Decavele M, Sonneville R, Beloncle F, Girault C, Dangers L, Lautrette A, Levrat Q, Rouze A, Vivier E, Lascarrou JB, Ricard JD, Razazi K, Barberet G, Lebert C, Ehrmann S, Massri A, Bourenne J, Pradel G, Bailly P, Terzi N, Dellamonica J, Lacave G, Robert R, Ragot S, Frat JP; HIGH-WEAN Study Group, for the REVA Research Network. Non-invasive ventilation alternating with high-flow nasal oxygen versus high-flow nasal oxygen alone after extubation in COPD patients: a post hoc analysis of a randomized controlled trial. Ann Intensive Care. 2021 Feb 9;11(1):30. doi: 10.1186/s13613-021-00823-7. PMID 33559765
- [Derived] Thille AW, Muller G, Gacouin A, Coudroy R, Decavele M, Sonneville R, Beloncle F, Girault C, Dangers L, Lautrette A, Cabasson S, Rouze A, Vivier E, Le Meur A, Ricard JD, Razazi K, Barberet G, Lebert C, Ehrmann S, Sabatier C, Bourenne J, Pradel G, Bailly P, Terzi N, Dellamonica J, Lacave G, Danin PE, Nanadoumgar H, Gibelin A, Zanre L, Deye N, Demoule A, Maamar A, Nay MA, Robert R, Ragot S, Frat JP; HIGH-WEAN Study Group and the REVA Research Network. Effect of Postextubation High-Flow Nasal Oxygen With Noninvasive Ventilation vs High-Flow Nasal Oxygen Alone on Reintubation Among Patients at High Risk of Extubation Failure: A Randomized Clinical Trial. JAMA. 2019 Oct 15;322(15):1465-1475. doi: 10.1001/jama.2019.14901. PMID 31577036
- [Derived] Thille AW, Muller G, Gacouin A, Coudroy R, Demoule A, Sonneville R, Beloncle F, Girault C, Dangers L, Lautrette A, Cabasson S, Rouze A, Vivier E, Le Meur A, Ricard JD, Razazi K, Barberet G, Lebert C, Ehrmann S, Picard W, Bourenne J, Pradel G, Bailly P, Terzi N, Buscot M, Lacave G, Danin PE, Nanadoumgar H, Gibelin A, Zanre L, Deye N, Ragot S, Frat JP; REVA research network. High-flow nasal cannula oxygen therapy alone or with non-invasive ventilation during the weaning period after extubation in ICU: the prospective randomised controlled HIGH-WEAN protocol. BMJ Open. 2018 Sep 5;8(9):e023772. doi: 10.1136/bmjopen-2018-023772. PMID 30185583